CLINICAL TRIAL: NCT01353625
Title: A Phase 1a/1b, Multicenter, Open Label, Dosefinding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the Dual Dna-pk and Tor Kinase Inhibitor, Cc-115, Administered Orally to Subjects With Advanced Solid Tumors and Hematologic Malignancies
Brief Title: Study to Assess Safety and Tolerability of Oral CC-115 for Patients With Advanced Solid Tumors, and Hematologic Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-115-ST-001
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Glioblastoma Multiforme; Squamous Cell Carcinoma of Head and Neck; Prostate Cancer; Ewing's Osteosarcoma; Chronic Lymphocytic Leukemia; Neoplasm Metastasis
Keywords: Neoplasm; Malignancy; Carcinoma; Lymphoma; Leukemia; Multiple myeloma; mTOR kinase inhibitor; Castration-resistant prostate cancer; Hormone-resistant prostate cancer; Diffuse Large B-cell lymphoma
MeSH Terms: conditions — Glioblastoma; Squamous Cell Carcinoma of Head and Neck; Prostatic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasm Metastasis; Neoplasms; Carcinoma; Lymphoma; Leukemia; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse | interventions — 1-ethyl-7-(2-methyl-6-(1H-1,2,4-triazol-3-yl)pyridin-3-yl)-3,4-dihydropyrazino(2,3-b)pyrazin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-115 (Experimental)
  Interventions: Drug: CC-115

INTERVENTIONS:
Drug: CC-115 — Part A (actively recruiting): Dose level starts with 0.5mg daily by mouth in cycles of 28 days. Level increases for different patient cohorts in 100% or 50% increments until optimal dose schedule is established for further study. Treatment continues for as long as patient benefits (i.e., until disease progression or unacceptable toxicity).
  Part B: Optimal dose schedule is administered in 28-day cycles until disease progression.

SUMMARY:
The main purpose of this first human study with CC-115 is to assess the safety and action of a new class of experimental drug (dual DNA-PK and TOR kinase inhibitors) in patients with advanced tumors unresponsive to standard therapies and to determine the appropriate dose and tumor types for later-stage clinical trials. The bioavailability of tablet and capsule formulations under fasting and fed conditions will also be evaluated in some patients.

DETAILED DESCRIPTION:
Latest amendment clarifies that Chronic Lymophocytic Leukemia (CLL) includes T-cell Prolymphocytic Leukemia (T-PLL). Prior treatment with some drugs targeting mTOR, P13K and related pathways is now permitted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed advanced solid tumor, chronic lymphocytic leukemia, small lymphocytic lymphoma, T-cell prolymphocytic leukemia, Non-Hodgkin Lymphoma or multiple myeloma
* Progressed or not tolerated standard therapy, and no further standard therapy is available
* Archival and screening tumor biopsy
* Eastern Cooperative Oncology Group Performance Status: 0 or 1
* Adequate organ function

Exclusion Criteria:

* Prior cancer-directed modalities or investigational drugs within 4 wks or 5 half lives, whichever is shorter
* Symptomatic brain metastases (prior treatment and stable metastases are allowed)
* Acute or chronic renal disease or pancreatitis
* Diarrhea ≥ Grade 2, impaired gastrointestinal absorption
* Impaired cardiac function
* History of diabetes requiring treatment, glucose >126 mg/dL, Glycated hemoglobin (HbA1c) ≥6.5%
* Peripheral neuropathy ≥ Grade 2
* Known Human Immunodeficiency Virus (HIV) infection, chronic hepatitis B or C (unless associated with hepatocellular cancer)
* Pregnant, inadequate contraception, breast feeding
* Most concurrent second malignancies
* Part B only: Prior treatment with agents targeting both mammalian target of rapamycin (mTOR) complexes (dual mammalian target of rapamycin complex 1/2 inhibitors) and/or PI3K/AKT pathways. However, prior treatment with isolated target of rapamycin complex 1 (TORC1) inhibitors (eg., rapalogs) is allowed in both parts of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-04-25 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | Continuously for 28 days after starting treatment
Non-Tolerated Dose | Continuously for 28 days after starting treatment
Maximum Tolerated Dose | Continuously for 28 days after starting treatment
Maximum Observed Concentration in Plasma of CC-115 | Days 1, 2, 15, 16 of treatment
Area Under the Concentration-Time Curve for CC-115 | Days 1, 2, 15 and 16 of treatment
Time to Maximum Concentration of CC-115 | Days 1, 2, 15, and 16 of treatment
Terminal Half-Life for CC-115 | Days 1, 2, 15, and 16 of treatment
Apparent Total Body Clearance of CC-115 | Days 1, 2, 15 and 16 of treatment
Apparent Volume of Distribution of CC-115 | Days 1, 2, 15, and 16 of treatment
Accumulation Index of CC-115 | Days 1, 2, 15 and 16 of treatment

SECONDARY OUTCOMES:
Pharmacodynamics | Screening (within 28 days prior to first dose of study drug) and Days 1, 2, 8, 15, 22, 28, 155, and end of treatment
  Phosphorylation inhibition determined by changes in the levels of multiple biomarkers including S6 and, 4EBP (for mTORC1), AKT (for mTORC2) and other appropriate biomarkers in circulating granulocytes and tumor tissue (when available).
Anti-Tumor Efficacy | Every 2-3 months until proof of tumor progression
  Tumor response rates using appropriate objective criteria for various malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of California, San Francisco Comprehensive Cancer Center and Cancer Research Institiute, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute Drug Development Unit, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Gustave Roussy, Villejuif, France
- Germany (2):
  - Uniklinik Koln, Cologne
  - Universitatsklinikum Wurzburg, Würzburg
- Spain (4):
  - Hospital Val d'Hebron, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital de Donosti, San Sebastián (Guipuzcoa)
  - Hospital Virgen del Rocio, Seville

REFERENCES:
- [Background] Thijssen R, Ter Burg J, Garrick B, van Bochove GG, Brown JR, Fernandes SM, Rodriguez MS, Michot JM, Hallek M, Eichhorst B, Reinhardt HC, Bendell J, Derks IA, van Kampen RJ, Hege K, Kersten MJ, Trowe T, Filvaroff EH, Eldering E, Kater AP. Dual TORK/DNA-PK inhibition blocks critical signaling pathways in chronic lymphocytic leukemia. Blood. 2016 Jul 28;128(4):574-83. doi: 10.1182/blood-2016-02-700328. Epub 2016 May 27. PMID 27235137
- [Derived] Munster P, Mita M, Mahipal A, Nemunaitis J, Massard C, Mikkelsen T, Cruz C, Paz-Ares L, Hidalgo M, Rathkopf D, Blumenschein G Jr, Smith DC, Eichhorst B, Cloughesy T, Filvaroff EH, Li S, Raymon H, de Haan H, Hege K, Bendell JC. First-In-Human Phase I Study Of A Dual mTOR Kinase And DNA-PK Inhibitor (CC-115) In Advanced Malignancy. Cancer Manag Res. 2019 Dec 13;11:10463-10476. doi: 10.2147/CMAR.S208720. eCollection 2019. PMID 31853198